CLINICAL TRIAL: NCT01117363
Title: Effect of Three Weeks Consumption of Rye Porridge Breakfast on 24 h Appetite Profile, and Acute Effect on OCTT and Breath Hydrogen
Brief Title: Effect of Three Weeks Consumption of Rye Porridge Breakfast
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Swedish University of Agricultural Sciences (Other)
Collaborators: Lantmannen Research and Development (Unknown); Good Food Practice, Sweden (Industry)
Responsible Party: Hanna Isaksson, Swedish University of Agricultural Sciences
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: SIV829
Record Dates: First submitted 2010-05-04; First posted 2010-05-05 (Estimated); Last update posted 2010-05-05 (Estimated); Status verified 2010-05

CONDITIONS: Obesity Prevention
Keywords: Appetite whole grain
MeSH Terms: interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rye porrige breakfast (Experimental)
  Interventions: Other: dietary intervention (rye porridge or wheat bread)
- Refined wheat reference bread breakfast (Active Comparator)
  Interventions: Other: dietary intervention (rye porridge or wheat bread)

INTERVENTIONS:
Other: dietary intervention (rye porridge or wheat bread) — A breakfast consisting of either active (rye porridge) or control (wheat bread) is given during 2 3-wk intervention periods in a randomized cross-over design. The two dietary intervention periods are separated by a 3-4 wks wash out.

SUMMARY:
Acute hunger-reducing effects (8h) has been documented for rye porridge breakfast compared with iso-caloric referenced refined wheat reference breakfast. The primary aim of the current study is to investigate whether this effects remains at regular consumption. A secondary aim is to compare the orocecal transit time (OCTT) between the two breakfasts.

DETAILED DESCRIPTION:
The study is randomised and cross-over. During two 3-wk periods, separated by a 3-4-wks wash out, subjects will consume test breakfasts. During one of the periods test breakfast includes rye flake porridge and during the other period test breakfast include bread made from sifted wheat. The breakfast meals will be similar in calorie-, protein-, carbohydrate- and fat content. For all other days but 1, 8 and 22 of respective test period, the breakfast foods will be handed out to the participants along with instructions to exchange their ordinary breakfast with the test foods. During day 1, 8 and 22 the breakfasts will be served at the study centre.

Following measurements will be made:

1. Subjective ratings of hunger, satiety and desire to eat during 24 h after breakfast on day 1, 8 and 22 during each 3-wk intervention period.
2. on day 8 during each intervention period, orocecal transit time and breath hydrogen will be measured after intake of the breakfast.
3. 3 day weighed food diaries will be taken at three occasions: at baseline and during the second week of each dietary intervention period.

ELIGIBILITY:
Inclusion Criteria:

* man or woman aged between 20 and 60 years;
* body mass index (BMI) 18-27 kg/m2;
* habit of consuming breakfast, lunch and dinner every day;
* and willingness to comply with the study procedures.

Exclusion Criteria:

* intake of medicine likely to affect appetite or food intake;
* any medical condition involving the gastrointestinal tract;
* eating disorder;
* smoking;
* consumption of more than three cups of coffee per day;
* change in body weight more than 10% during three months prior to screening;
* consumption of any restricted diet such as vegan, gluten-free, slimming;
* pregnancy, lactation or wish to become pregnant during the study period;
* any known intolerance towards salazopyrin and similar substances

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2010-03; Primary Completion 2010-07 (Estimated); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
Appetite profile | 24 h
  Subjective feelings of appetite (hunger, satiety and desire to eat) were assessed every 30 min, starting just before breakfast at 08:00 and continuing until bedtime. The last recording was made before breakfast on the following day.

SECONDARY OUTCOMES:
energy intake | 3 days
  Weighed food records was completed by the subjects during baseline and each intervention phase.
Orocecal transit time | 8 h
  Salazopyrin (two 500 mg tabelts) is taken after breakfast. The substance passes the stomach and small intestine unabsorbed and is broken down by microbial fermentation in the colon to sulphapyridine and 5-ASA. Sulphapyridine appearance in the blood is then measured as an indicator of colon arrival time.
Breath hydrogen | 8 h

CONTACTS AND LOCATIONS:
Overall Officials: Per Åman, Professor, Study Director — Swedish University of Agricultural Sciences
Locations (1):
- Good Food Practice, Uppsala, Sweden

REFERENCES:
- [Derived] Isaksson H, Tillander I, Andersson R, Olsson J, Fredriksson H, Webb DL, Aman P. Whole grain rye breakfast - sustained satiety during three weeks of regular consumption. Physiol Behav. 2012 Feb 1;105(3):877-84. doi: 10.1016/j.physbeh.2011.10.023. Epub 2011 Oct 28. PMID 22061429